CLINICAL TRIAL: NCT01080027
Title: An International, Multi Centre, Prospective, Observational Study of Safety, Tolerability and Adherence of Patients With Relapsing Remitting Multiple Sclerosis Administered Interferon Beta-1a (Rebif® New Formulation) in Real Life Settings
Brief Title: Safety, Tolerability and Adherence With Rebif® New Formulation in Real Life Settings (STAR)
Acronym: STAR
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck A.E., Greece (Industry); Merck OY, Finland (Industry); Merck B.V., Netherlands (Industry); Merck A.B., Sweden (Industry); Merck, S.A., Portugal (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 701068_506
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis, Relapsing Remitting
Keywords: Multiple sclerosis; Relapsing remitting; Rebif
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Rebif® New Formulation — The recommended dose of Rebif® is 22 or 44 μg administered three times per week by subcutaneous injection.
  Other Names: Interferon beta1-A

SUMMARY:
The rationale of this study is to assess the safety profile, efficacy and adherence to Rebif® New Formulation in real life settings with a multinational approach, as well as the impact of this improved formulation (with regards to adverse events [AEs]) to subjects' adherence.

DETAILED DESCRIPTION:
This international, multicentric, prospective, observational study is being conducted to assess the safety profile, efficacy and adherence to Rebif® New Formulation in real life settings in subjects with relapsing remitting multiple sclerosis (RRMS), as well as the impact of this improved formulation (with regards to adverse events [AEs]) to subjects' adherence. Three hundred and fifty subjects from approximately 80 sites across seven countries will be enrolled in the study. Subjects will be treated with IFN beta-1a (Rebif® New Formulation) in real life settings according to the clinical and paraclinical course and laboratory findings as routinely evaluated by the physician. Data related to AEs; subjects' adherence to treatment, reasons for treatment discontinuation; number and reasons of missed injections; and the clinical and paraclinical data on efficacy regarding relapses will be captured. Data will be reported prospectively throughout the duration of the study (12 months) at two visits (at month 6 and month 12) following the initial visit; at baseline, data can be recorded retrospectively from the subjects' medical file. All the data will be evaluated descriptively.

OBJECTIVES

Primary objective

* To assess the local tolerability of Rebif® New Formulation in real life settings with a multinational approach.

Secondary objectives

* To assess the safety profile, subjects' adherence to and efficacy of Rebif® New Formulation

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of RRMS according to the Mc Donald criteria(2005)
* 18 to 60 years of age
* Expanded Disability Status Scale (EDSS) < 6
* Naïve subjects or subjects treated with Rebif® New Formulation for no more than 6 weeks prior to enrollment
* Subjects who have given written informed consent to participate in the study

Exclusion Criteria:

* Primary progressive or secondary progressive MS
* Subjects previously administered IFN beta-1a (including Rebif®) or IFN beta-1b or glatiramer acetate or any other immunomodulatory or immunosuppressive agents or any other MS therapy in the past with the exception of Rebif® New Formulation for no more than 6 weeks prior to enrollment
* Subjects receiving oral or systemic corticosteroids or Adrenocorticotrophic hormone within 30 days of visit 1 (prior to enrolment)
* History of any chronic pain syndrome
* Known allergy to IFN or its excipients
* Serious or acute heart disease such as uncontrolled cardiac dysrhythmias, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure
* Inadequate liver function, defined by a alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN), or alkaline phosphatase > 2 x ULN, or total bilirubin > 2 x ULN if associated with any elevation of ALT or alkaline phosphatase
* Inadequate bone marrow reserve, defined as a white blood cell count less than 0.5 x lower limit of normal
* Current or past (within the last 2 years) history of alcohol or drug abuse
* Contra-indications to IFN beta-1a

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects diagnsoed with RRMS from approximately 80 sites across seven countries.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with injection site reactions (ISRs) | Baseline, month 6 and month 12

SECONDARY OUTCOMES:
proportion of subjects with AEs and with specific categories of AEs; proportion and reasons of missed injections, annual relapse rate, proportion of relapse-free subjects from baseline, time to first relapse | Baseline, month 6 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Michalis Arvanitis, MD, MSc, Study Director — Merck A.E., Greece
Locations (1):
- Neurology Clinic, General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki, Greece

REFERENCES:
- [Derived] Hupperts R, Ghazi-Visser L, Martins Silva A, Arvanitis M, Kuusisto H, Marhardt K, Vlaikidis N; STAR Study Group. The STAR Study: a real-world, international, observational study of the safety and tolerability of, and adherence to, serum-free subcutaneous interferon beta-1a in patients with relapsing multiple sclerosis. Clin Ther. 2014 Dec 1;36(12):1946-1957. doi: 10.1016/j.clinthera.2014.04.002. Epub 2014 May 5. PMID 24811754